CLINICAL TRIAL: NCT04187456
Title: An Open Label, 2 Period, Fixed-sequence Study to Assess the Effect of Savolitinib on the Pharmacokinetics of Oral Midazolam (a CYP450 3A Probe) in Healthy Subjects
Brief Title: A Study in Healthy Male Subjects to Understand How Savolitinib When Taken With Midazolam Behaves Inside the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D5084C00004
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumors
Keywords: Pharmacokinetics; Safety; Small molecule kinase inhibitor; Open-label
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam + Savolitinib (Experimental): * Treatment Period 1: Single administration of midazolam (1 mg) will occur on Study Day 1, after a high fat, high calorie breakfast, followed by PK sampling for 24 hours.
  * Treatment Period 2: Single administration of midazolam 1 mg in combination with a single administration of savolitinib (600 mg), after a high fat, high calorie breakfast will occur on Study Day 5 and PK sampling will occur for 24 hours.
  Interventions: Drug: Savolitinib; Drug: Midazolam

INTERVENTIONS:
Drug: Savolitinib — Single dose (together with midazolam) on Study Day 5 after a high fat, high calorie breakfast.
Drug: Midazolam — Single dose (alone) on Study Day 1 and single dose (together with savolitinib) on Study Day 5, both after a high fat, high calorie breakfast.

SUMMARY:
This study will be an open label, 2 period, fixed sequence study in healthy male subjects, performed at a single study center in the Unites States of America. The purpose of this study is to evaluate the effect of savolitinib on the PK of midazolam, a known cytochrome P450 (CYP) 3A substrate.

DETAILED DESCRIPTION:
This study is designed as an open-label, 2 treatment period, fixed sequence study in healthy male subjects, performed at a single study center.

The study will comprise:

* A screening period of maximum 28 days;
* Two treatment periods:

Treatment Period 1 consists of 5 days (Study Days -1 to 4), starting with admission to the Study Center on Study Day -1, dosing of midazolam alone on Study Day 1 and ending on Study Day 4, after a 3 day washout period.

Treatment Period 2 consists of 2 days (Study Days 5 and 6), with administration of midazolam in combination with savolitinib on Study Day 5. Subjects will be discharged from the Study Center on Study Day 6, after the last PK sample is collected.

* The Follow up Visit will occur at least 14 days (Study Day 19 or after) after the administration of savolitinib in Treatment Period 2.
* Subjects will be admitted to the Study Center on Study Day -1, prior to the evening meal the night before dosing with midazolam alone (Study Day 1) and will stay in house until at least 24 hours after dosing with midazolam in combination with savolitinib (Study Day 5). Subjects will thus be discharged on Study Day 6, after the last PK sample has been collected.

Each subject will be involved in the study between 21 and approximately 48 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects, aged 18 - 65 years (inclusive) , with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 35 kg/m2 inclusive and body weight greater than 50 kg and no more than 100 kg.
4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and Total Bilirubin (TBL) less than or equal to upper limit of normal for the institution at screening.
5. Have a calculated creatinine clearance (CrCL) greater than 80 mL/min using the Cockcroft-Gault formula at screening.
6. Provision of a signed, written and dated informed consent for optional genetic/biomarker research. If a subject decline to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in the protocol..

Exclusion Criteria:

1. Healthy subjects of Japanese ethnicity and any healthy subject that has 1 parent or grandparent (maternal or paternal) of Japanese ethnicity.
2. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
3. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
5. Planned in-patient surgery, dental procedure or hospitalizing during the study.
6. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the PI.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
8. Abnormal vital signs, after 5 minutes supine rest, defined as any of the following:

(1) Systolic BP < 90 mmHg or ≥ 140 mmHg (2) Diastolic BP < 50 mmHg or ≥ 90 mmHg (3) Heart rate < 45 or > 85 beats per minute. 9 Any clinically significant abnormalities in rhythm, conduction or morphology of the 12-lead resting ECG that may interfere with the interpretation of QTc interval changes.

These include healthy subjects with any of the following:

1. Abnormal ST-T-wave morphology, particularly in the protocol defined primary lead (V2) or left ventricular hypertrophy.
2. PR interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
3. PR interval prolongation (> 200 ms). Intermittent second (Type 1 second degree block [Wenckebach Phenomenon] while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
4. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
5. Mean resting correct QT interval (QTcF) > 450 ms for men on screening obtained from 3 ECGs or history or factors that may increase the risk of QTcF prolongation such as chronic hypokalemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes (TdP).

10 Known or suspected history of drug abuse, as judged by the Principal Investigator.

11 Current smokers or those who have smoked or used nicotine products within the previous 30 days.

12 History of alcohol abuse, as judged by the PI, or excessive intake of alcohol (defined as an average weekly intake of > 21 units or an average daily intake of > 3 units).

13 Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator.

14 Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the administration of IMP.

15 Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the firs admission on Day -1.

16 Use of any prescribed or non-prescribed medication including antacids, analgesics (other than use of ibuprofen) up to 72 hours before first dosing day until final follow-up visit, herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer (5 times half-life) if the medication has a long half-life.

17 Positive screen for drugs of abuse, cotinine (nicotine) and/or alcohol at screening and at admission to the Study Center and/or positive screen for alcohol on admission to the Study Center (Day -1, Treatment Period 1).

18 History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib or midazolam.

19 Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.

20 Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit, whichever is the longest.

Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.

21 Known or suspected history of alcohol abuse or excessive intake of alcohol as judged by the PI.

22 Involvement of any AstraZeneca, Parexel or study site employee or their close relatives.

23 Subjects who have previously received savolitinib or midazolam. 24 Judgement by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

25 Subjects who are vegans, vegetarians or have medical dietary restrictions and who are lactose intolerant.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Midazolam: Area under the plasma concentration-time curve from time zero to infinity (AUC) ratio of geometric means of test treatment (midazolam + savolitinib), relative to reference treatment (midazolam alone). | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To assess the effect of savolitinib on the PK of midazolam.
Midazolam: Maximum observed plasma concentration (Cmax) ratio of geometric means of test treatment (midazolam + savolitinib), relative to reference treatment (midazolam alone). | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To assess the effect of savolitinib on the PK of midazolam.

SECONDARY OUTCOMES:
Midazolam: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-t)] ratios of geometric means of test treatment (midazolam + savolitinib), relative to reference treatment (midazolam alone). | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam: Cmax | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam: [AUC(0-t)] | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam: Time to reach maximum observed plasma concentration (tmax) | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration time curve (t½,λz) | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam: Terminal elimination rate constant (λz) | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam and savolitinib: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Midazolam and savolitinib: Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Treatment period 1 and 2 (Study Days 1,2, 5 and 6). Midazolam- pre dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose on Study Days 1 and 5. Savolitinib- pre-dose and 1,2, 4, 6, 8, 12 and 24 hours post dose.
  To describe the PK of midazolam in the presence and absence of savolitinib.
Number of subjects with adverse events | At screening, Day -1, 1, 2, 3, 4, 5, 6, 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal systolic blood pressure (BP) | At screening, Day -1, 1, 2, 5, 6, 19. Vital signs on dosing days will be collected at pre dose, 0.5, 1, 2, 3, 4, 8 and 24 hours post dose.
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal diastolic blood pressure (BP) | At screening, Day -1, 1, 2, 5, 6, 19. Vital signs on dosing days will be collected at pre dose, 0.5, 1, 2, 3, 4, 8 and 24 hours post dose.
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in pulse rate | At screening, Day -1, 1, 2, 5, 6, 19. Vital signs on dosing days will be collected at pre dose, 0.5, 1, 2, 3, 4, 8 and 24 hours post dose.
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in physical examination | At screening, Day -1, 1, 2, 3, 4, 5, 6 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in White blood cell (WBC) count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Red blood cell (RBC) count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Hemoglobin (Hb) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Hematocrit (HCT) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Mean corpuscular volume (MCV) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Mean corpuscular hemoglobin (MCH) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Mean corpuscular hemoglobin concentration (MCHC) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Neutrophils absolute count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Monocytes absolute count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Eosinophils absolute count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Basophils absolute count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Platelets | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Reticulocytes absolute count | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in sodium | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in pottasium | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in urea | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in creatinine | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in albumin | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in calcium | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in phosphate | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in glucose (fasting) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in C-reactive protein (CRP) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in T4 | At screening
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Thyroid-Stimulating Hormone (TSH) | At screening
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Alkaline phosphatase (ALP) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Alanine aminotransferase (ALT) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Aspartate aminotransferase (AST) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in Gamma glutamyl transpeptidase (GGT) | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in total bilirubin | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in unconjugated bilirubin | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in urinalysis | At screening, Day 1, 4, 5 and 19
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.
Number of subjects with abnormal findings in pulse oximetry | Day 1 and 5
  To examine the safety and tolerability of midazolam alone and in combination with savolitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States